CLINICAL TRIAL: NCT00388557
Title: Effect of Ketoconazole on the Pharmacokinetics of Intravenous (IV) Vinflunine in Patients With Advanced Cancer
Brief Title: Effect of Ketoconazole on the Pharmacokinetics of Vinflunine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA183-009
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: vinflunine + ketaconazole

INTERVENTIONS:
Drug: vinflunine + ketaconazole — vinflunine solution for injection, ketaconazole tablets, vinflunine IV, ketaconazole oral, vinflunine 80 to 320mg/m2 + ketaconazole 400 mg, vinflunine every 3 wks, ketaconazole C1 only, variable duration

SUMMARY:
The purpose of the study is to test how ketoconazole affects with handling of vinflunine by the body which might affect how much vinflunine is in the blood stream and for how long

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer excluding cancer within the blood, adequate kidney and liver function.

Exclusion Criteria:

* Prior use of vinflunine, other active medical disorders, severe nerve damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the effect of ketoconazole on the pharmacokinetics of vinflunine in patient with advanced cancer. A total of 28 blood samples will be collected | Days 1 through 5 and Day 8 of Cycles 1 and 2

SECONDARY OUTCOMES:
Evaluate the safety of vinflunine co-administered with ketoconazole and assess the safety of vinflunine in patients with advanced cancer. Safety laboratory assessments and evaluations will be collected | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Tennessee Oncology, Pllc, Nashville, Tennessee, United States